CLINICAL TRIAL: NCT00866307
Title: Intensified PEG-Asparaginase in High Risk Acute Lymphoblastic Leukemia (ALL): A Pilot Study
Brief Title: Pegaspargase and Combination Chemotherapy in Treating Younger Patients With Newly Diagnosed High-Risk Acute Lymphoblastic Leukemia (Closed to Accrual 4-22-2011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL08P1; NCI-2009-01169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000636174; COG-AALL08P1; AALL08P1 (Other: Children's Oncology Group); AALL08P1 (Other: CTEP); U10CA098413 (NIH); U10CA180886 (NIH); U10CA180899 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia; Childhood B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisone; deltacortene; prednylidene; Thioguanine; Vincristine

ARMS (2):
- Arm I (HR-average) (Experimental): See Detailed Description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm II (HR-high) (Experimental): See Detailed Description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Radiation: Prophylactic Cranial Irradiation; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT and IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: Arm II (HR-high)
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT and PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given IV or PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
  Arms: Arm II (HR-high)
Radiation: Prophylactic Cranial Irradiation — Undergo radiation
  Other Names: PCI
  Arms: Arm II (HR-high)
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This pilot clinical trial studies the side effects of pegaspargase when given together with combination chemotherapy in treating patients with newly diagnosed high-risk acute lymphoblastic leukemia. Pegaspargase may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) together with pegaspargase may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that biweekly intravenous (IV) pegaspargase beginning with Consolidation and ending with completion of delayed intensification (DI) in combination with hemi-augmented BFM therapy (hABFM) is feasible and safe in children with high risk (HR) acute lymphoblastic leukemia (ALL).

OUTLINE: Patients are stratified according to risk assignment (high-risk [HR]-average [day 29 minimal residual disease (MRD) < 0.01%] vs HR-high [MRD >= 0.01%, presence of central nervous system [CNS]3 leukemia, testicular disease, myeloid/mixed lineage leukemia [MLL] rearrangement, hypodiploidy, or steroid therapy within the past month]). Patients are assigned to 1 of 2 treatment groups.*

(Note: *Amendment 2 [4-22-2011] requires changes in the regimens. See the changes below, after Maintenance therapy.)

INDUCTION THERAPY: All patients receive cytarabine intrathecally (IT) on day 1; vincristine sulfate IV on days 1, 8, 15, and 22; prednisone IV or orally (PO) twice daily (BID) on days 1-28; daunorubicin hydrochloride IV over 15 minutes on days 1, 8, 15, and 22; methotrexate IT on days 8 and 29*; and pegaspargase IV over 1-2 hours on day 4.

(Note: *Patients with CNS3 disease [white blood cells [(WBC)] >= 5/uL and positive for blasts on cytospin] also receive methotrexate IT on days 15 and 22.)

CONSOLIDATION THERAPY (begins on day 36 of induction therapy):

GROUP A (HR-AVERAGE): Patients receive cyclophosphamide IV over 1 hour on days 1 and 29; cytarabine IV over 15 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO once daily (QD) on days 1-14 and 29-42; vincristine sulfate IV on days 15, 22, 43, and 50; methotrexate IT on days 1, 8, 15*, and 22*; and pegaspargase IV over 1-2 hours on days 15 and 43.

GROUP B (HR-HIGH): Patients receive cyclophosphamide, cytarabine, mercaptopurine, vincristine sulfate, and methotrexate as in Group A. Beginning on day 1, patients also receive pegaspargase IV over 1-2 hours every 2 weeks. Patients with CNS3 disease undergo cranial radiotherapy QD for 10 days and patients with testicular disease undergo testicular radiotherapy QD for 12 days, beginning on day 1 of consolidation.

(Note: *Patients with CNS3 disease [WBC >= 5/uL and positive for blasts on cytospin] do not receive methotrexate IT on days 15 and 22.)

Interim maintenance (IM) therapy (begins on day 57 of consolidation):

GROUP A: Patients receive vincristine sulfate IV on days 1, 11, 21, 31, and 41; methotrexate IV over 10-15 minutes on days 1, 11, 21, 31, and 41; methotrexate IT on days 1 and 31; and pegaspargase IV over 1-2 hours on days 2 and 22.

GROUP B: Patients receive vincristine sulfate and methotrexate as in Group A. Beginning on day 1, patients also receive pegaspargase IV over 1-2 hours every 2 weeks.

DI therapy (begins on day 57 of IM):

GROUP A: Patients receive vincristine sulfate IV on days 1, 8, 15, 43, and 50; dexamethasone IV or PO BID on days 1-7 and 15-21; doxorubicin hydrochloride IV over 15 minutes on days 1, 8, and 15; cyclophosphamide IV over 1 hour on day 29; cytarabine IV over 15 minutes or SC on days 29-32 and 36-39; thioguanine PO on days 29-42; methotrexate IT on days 1, 29, and 36; and pegaspargase IV over 1-2 hours on days 4 and 43.

GROUP B: Patients receive vincristine sulfate, dexamethasone, doxorubicin hydrochloride, cyclophosphamide, cytarabine, thioguanine, and methotrexate as in Group A. Beginning on day 1, patients also receive pegaspargase IV over 1-2 hours every 2 weeks.

MAINTENANCE THERAPY (MT; begins on day 57 of DI): All patients receive vincristine sulfate IV on days 1, 29, and 57; prednisone PO BID on days 1-5, 29-33, and 57-61; mercaptopurine PO on days 1-84; methotrexate IT on day 1; and methotrexate PO BID on days 8, 15, 22, 29*, 36, 43, 50, 57, 64, 71, and 78.

In both groups, MT repeats every 12 weeks until total duration of therapy is 2 years from the start of IM for female patients and 3 years from the start of IM for male patients. Patients in Group B who did not undergo radiotherapy to the brain during consolidation therapy undergo prophylactic cranial radiotherapy (CR) daily for 8 days.

([Note: *Patients in Group A also receive methotrexate IT on day 29 of courses 1-4 [no oral methotrexate]).

REVISED MT (RMT): The regimen is the same as standard MT, but 2 of the doses of IT methotrexate are omitted (day 29 of courses 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be eligible for and enrolled on AALL03B1 or the successor classification study
* Patients must have newly diagnosed high-risk B-precursor acute lymphoblastic leukemia (ALL)
* WBC criteria

  * Age 1.00-9.99 years: WBC >= 50,000/uL
  * Age 10.00 - 30.99 years: Any WBC
  * Prior steroid therapy: Any WBC
  * Patients with testicular leukemia: Any WBC
* Patients shall have had no prior cytotoxic chemotherapy with the exception of steroids and intrathecal cytarabine
* Intrathecal chemotherapy with cytarabine is allowed prior to registration for patient convenience; this is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture; the CNS status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment; systemic chemotherapy must begin within 72 hours of this intrathecal therapy
* Patients receiving prior steroid therapy are eligible for study; the dose and duration of previous steroid therapy should be carefully documented
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Pregnant female patients are ineligible; pregnancy tests with a negative result must be obtained in all post-menarchal females; males and females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method; lactating females must agree that they will not breastfeed a child while on this study
* Patients with Down syndrome (DS) are ineligible since excessive toxicities and death have been noted for those enrolled on AALL0232 receiving the prednisone/Capizzi methotrexate (PC) arm of treatment, which is the backbone regimen for the current study

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 104 (Actual)
Dates: Start 2009-02-23 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ZoAnn E Dreyer, Principal Investigator — Children's Oncology Group
Locations (28):
- United States (25):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
- Australia (2):
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with newly diagnosed high-risk B-precursor acute lymphoblastic leukemia (ALL), no prior cytotoxic chemotherapy besides steroids and intrathecal cytarabine and WBC criteria: Age 1.00-9.99 years: WBC >= 50,000/uL; Age 10.00 - 30.99 years or prior steroid therapy or with testicular leukemia: Any WBC
Pre-assignment Details: Patients with Day 29 Marrow counts >25% (M3) or pegaspargase contraindication go off therapy before risk stratification.
Groups:
- Induction: All Patients
- Group A (High Risk-Average): Patients with day 29 MRD <0.01% and no CNS3, testicular disease, steroid pretreatment, MLL+, or hypodiploidy. Treated with Standard PEG-asparaginase therapy (hABFM)
- Group B (High Risk-High): Patients with day 29 MRD >=0.01% or at least one of: CNS3, Testicular disease, Steroid Pre-treatment, MLL+, or hypodiploidy. Received Intensified PEG-asparaginase therapy
Period: Induction
Arm/Group | Induction | Group A (High Risk-Average) | Group B (High Risk-High)
Started | 104 | 0 | 0
Completed | 84 | 0 | 0
Not Completed | 20 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Identification of Patients with Day 29 M | 3 | 0 | 0
Not completed — Inadequate cytognetic samples th | 1 | 0 | 0
Not completed — Improper post-induction consent | 2 | 0 | 0
Not completed — Study was closed at the time | 1 | 0 | 0
Period: Consolidation/Maintenance
Arm/Group | Induction | Group A (High Risk-Average) | Group B (High Risk-High)
Started | 0 | 54 | 30
Completed | 0 | 45 | 14
Not Completed | 0 | 9 | 16
Not completed — Adverse Event | 0 | 0 | 8
Not completed — Death | 0 | 0 | 1
Not completed — Physician Decision | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Development of 2nd malignant neoplasm | 0 | 0 | 2
Not completed — Recurrent leukemia following remission | 0 | 3 | 1
Not completed — Therapy error | 0 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Patient moved to non-participating inst | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction
Number analyzed (Participants) | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 96
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 7
  White | 68
  More than one race | 0
  Unknown or Not Reported | 21

OUTCOME MEASURES:

1. Primary Outcome: AALL08P1 Safety Outcome
Description: Percentage of Group B (High Risk-High) patients taking less than 49 weeks from day 1 of consolidation to day 1 of maintenance therapy. Only Group B analyzed since this is prespecified in protocol.
Time Frame: Consolidation through Delayed Intensification
Population: Patients with High Risk-High (Group B) Acute Lymphoblastic Leukemia (ALL)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Group B (High Risk-High)
Number analyzed (Participants) | 30
percentage of participants | 50.0 [35.6 to 64.4]
Statistical Analysis 1: Comparison: Group B (High Risk-High); Per protocol, percentage of high risk-High patients taking less than 49 weeks from day 1 of consolidation to day 1 of maintenance therapy is compared to a null fixed rate (<=73%). A 90% two-sided Agresti-Coull confidence interval will be constructed and the lower bound examined. Will reject null if lower bound of confidence interval is above 73%; Test type: Superiority or Other; Agresti-Coull Confidence Interval; Percentage = 50.0, 90% CI 2-sided [35.6 to 64.4]

2. Primary Outcome: AALL08P1 Feasibility Outcome
Description: Percentage of Group B (High Risk-High) patients that tolerate at least 8 of the 12-14 total doses of pegaspargase during Consolidation, Interim Maintenance, and Delayed Intensification periods. Only Grp B analyzed since this is prespecified in protocol.
Time Frame: Consolidation through Delayed Intensification
Population: Patients with High Risk-high Acute Lymphoblastic Leukemia (ALL)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Group B (High Risk-High)
Number analyzed (Participants) | 30
percentage of participants | 53.3 [38.7 to 67.4]
Statistical Analysis 1: Comparison: Group B (High Risk-High); Per protocol, percentage receiving at least 8 doses is compared to a null fixed rate (<=42%). A 90% two-sided Agresti-Coull confidence interval will be constructed. Will reject null if lower bound of confidence interval is above 42%; Test type: Superiority or Other; Agresti-Coull Confidence Interval; Percentage = 53.3, 90% CI 2-sided [38.7 to 67.4]

ADVERSE EVENTS:
Arm/Group | Induction | Group A (High Risk-Average) | Group B (High Risk-High)
Serious Adverse Events (participants affected / at risk) | 10/104 | 1/54 | 4/30
Other Adverse Events (participants affected / at risk) | 97/104 | 53/54 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (N=104) | Group A (High Risk-Average) (N=54) | Group B (High Risk-High) (N=30)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (6) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (N=104) | Group A (High Risk-Average) (N=54) | Group B (High Risk-High) (N=30)
Abdominal infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 8 (9) | 3 (3)
Abducens nerve disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 2 (3) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 47 (100) | 28 (70) | 15 (25)
Alkaline phosphatase increased (Investigations) | 4 (4) | 3 (3) | 1 (1)
Allergic reaction (Immune system disorders) | 10 (11) | 7 (8) | 3 (3)
Anaphylaxis (Immune system disorders) | 15 (17) | 9 (11) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 32 (58) | 18 (35) | 11 (19)
Anorectal infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 7 (8) | 3 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (3) | 2 (3) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Arachnoiditis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 23 (30) | 14 (20) | 7 (8)
Ataxia (Nervous system disorders) | 2 (3) | 2 (3) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 9 (22) | 7 (19) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 19 (29) | 10 (15) | 6 (11)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 6 (8) | 6 (8) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 57 (130) | 38 (85) | 18 (44)
Fever (General disorders) | 5 (5) | 4 (4) | 0 (0)
Fibrinogen decreased (Investigations) | 11 (15) | 7 (11) | 3 (3)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 1 (1)
GGT increased (Investigations) | 9 (9) | 1 (1) | 6 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 5 (6) | 4 (5) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 3 (4) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 24 (31) | 12 (18) | 8 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (8) | 4 (4) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 7 (7) | 2 (2) | 4 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (12) | 3 (3) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (12) | 7 (8) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 12 (16) | 6 (8) | 4 (6)
Hyponatremia (Metabolism and nutrition disorders) | 20 (24) | 10 (13) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 3 (3) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 4 (8) | 3 (7) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 62 (155) | 39 (98) | 17 (39)
Infective myositis (Infections and infestations) | 1 (2) | 1 (2) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 1 (1)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 4 (4) | 3 (3) | 1 (1)
Lipase increased (Investigations) | 10 (13) | 5 (8) | 3 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 10 (16) | 7 (11) | 3 (5)
Lymph gland infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (4) | 2 (4) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 10 (10) | 6 (6) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3 (7) | 1 (4) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (4) | 1 (2) | 1 (2)
Neutrophil count decreased (Investigations) | 72 (212) | 47 (144) | 21 (61)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Oculomotor nerve disorder (Nervous system disorders) | 2 (3) | 1 (2) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Pain (General disorders) | 4 (4) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (13) | 5 (6) | 3 (3)
Pancreatic enzymes decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 7 (9) | 4 (6) | 2 (2)
Papilledema (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 20 (30) | 10 (13) | 9 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 22 (31) | 13 (16) | 7 (12)
Personality change (Psychiatric disorders) | 3 (4) | 2 (2) | 1 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 34 (70) | 20 (37) | 11 (22)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 5 (5) | 4 (4) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 5 (6) | 3 (4) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4) | 0 (0)
Skin infection (Infections and infestations) | 5 (6) | 2 (2) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue necrosis upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 6 (7) | 3 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (9) | 3 (4) | 1 (5)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 8 (11) | 6 (9) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight loss (Investigations) | 6 (8) | 4 (5) | 2 (3)
White blood cell decreased (Investigations) | 37 (102) | 22 (64) | 12 (33)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The COG SDC reviewed the NLM notification related to ct.gov AE/SAE reporting. The information in 'Additional Description' is accurate with respect to data supplied to ct.gov.COG plans to submit data AE/SAE data consistent with the text in this field.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.